CLINICAL TRIAL: NCT01636804
Title: Incidence & Predictors of Mechanical Abnormalities of QuickSite® and QuickFlex® Left Ventricular Pacing Leads: Impact on Electrophysiological Profile
Brief Title: Incidence & Predictors of Mechanical Abnormalities of QuickSite® and QuickFlex® Left Ventricular Pacing Leads
Status: Completed | Type: Observational
Sponsor: Dhanunjaya Lakkireddy, MD, FACC (Other)
Responsible Party: Sponsor-Investigator, Dhanunjaya Lakkireddy, MD, FACC, Associate Professor, University of Kansas Medical Center
Organization: University of Kansas Medical Center (Other)
Other Study IDs: 13211
Record Dates: First submitted 2012-07-05; First posted 2012-07-10 (Estimated); Last update posted 2013-08-09 (Estimated); Status verified 2013-08

CONDITIONS: Left Ventricular Pacing Leads
Keywords: Quicksite; Quickflex; St. Jude Medical

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Quicksite and Quickflex: Patients who have received the leads affected by the medical product advisory
  Interventions: Device: Quicksite; Device: Quickflex

INTERVENTIONS:
Device: Quicksite — St. Jude Medical produced lead called Quicksite
Device: Quickflex — St. Jude Medical produced lead called Quickflex

SUMMARY:
On April 2, 2012 the manufacturer of the Quicksite® and Quickflex® leads, St. Jude Medical, released a voluntary medical device advisory regarding these leads' potential for problems with the silicone insulation covering one end of the lead, where it meets another section of the lead which is coated with a different insulating material (polyurethane). There has been a voluntary suspension of sales of these leads.

There are approximately 179,000 of the above leads implanted worldwide with an estimated 101,000 leads currently in service (59,000 in US). There have been 39 confirmed cases of the conductor portion of the lead becoming exposed from the silicone insulation (externalization), and the rate of occurrence of this type of problem is conservatively estimated at less than one percent. However, a review done by St. Jude Medical of returned Quicksite® and Quickflex® leads and available X-ray and fluoroscopic (x-ray movie) images of patients with these leads (from 1,219 patients) revealed a higher rate of 3-4%. It is presumed that there are patients whose leads have not yet been affected by this problem, but whose leads may show signs of structural changes on x-ray or fluoroscopy. This study seeks to determine what structural changes may be occurring in these leads, what signs might predict these changes, and what impact these changes may have on the lead and its performance.

ELIGIBILITY:
Inclusion Criteria:

* Patient that received Quicksite or Quickflex lead at the University of Kansas Hospital

Exclusion Criteria:

* Not willing to consent to data collection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients that received either Quicksite or Quickflex leads at the University of Kansas Hospital
Sampling Method: Non-Probability Sample
Enrollment: 190 (Estimated)
Dates: Start 2012-07

PRIMARY OUTCOMES:
Evaluate the mechanical/structural abnormalities in implanted St Jude Medical QuickSite® and QuickFlex® left ventricular (LV) pacing leads

CONTACTS AND LOCATIONS:
Overall Officials: Dhanunjaya Lakkireddy, MD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States